CLINICAL TRIAL: NCT04937855
Title: The Mechanism of lncRNA NEAT1 in Alleviating Acute Respiratory Distress Syndrome Through miR-27b Regulated Nrf2 Pathway
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Guangfa Zhu, Director, Head of Respiratory and Critical Medicine Department, Beijing Anzhen Hospital
Other Study IDs: 81970067
Record Dates: First submitted 2020-01-11; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Acute Respiratory Distress Syndrome; Inflammation
Keywords: long non-coding RNA NEAT1; microRNA-27b; nuclear factor E2-related factor 2
MeSH Terms: conditions — Respiratory Distress Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and BALF will be stored at -70˚C
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control group: 25 gender and age matching healthy controls
  Interventions: Other: no intervention
- ARDS group 1: 100 ARDS patients at the time of check in hospital
  Interventions: Other: no intervention
- ARDS group 2: 100 ARDS patients at the time of 24h after check in hospital
  Interventions: Other: no intervention
- ARDS group 3: 100 ARDS patients at the time of 48h after check in hospital
  Interventions: Other: no intervention
- ARDS group 4: 100 ARDS patients at the time of 72h after check in hospital
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
The acute respiratory distress syndrome, formerly known as the acute lung injury (ARDS/ALI), is a critical illness with high mortality due to the lack of effective treatment. The pathogenesis of ARDS/ALI has not been fully elucidated. Nuclear factor E2-related factor 2 (Nrf2) plays a key role in regulating lung inflammation and oxidative stress which are closely related to lung injury in ARDS/ALI, but its regulatory mechanism remains unclear. The investigator's provious study shown that microRNA-27b (miR-27b) downregulated Nrf2 to aggravate lung inflammation and histological injury. Furthermore, in lipopolysaccharide (LPS)-induced cell (J774A.1) inflammation model, miR-27b was upregulated while the long non-coding RNA (lncRNA) NEAT1 was downregulated, the putative binding sites of lncRNA NEAT1 and miR-27b were successfully predicted by bioinformatics approach. Thus, the investigators propose that NEAT1 plays as a competing endogenous RNA (ceRNA) to adsorb miR-27b and liberate Nrf2, therefore, to attenuate lung inflammation and related lung injury in ARDS/ALI. This project aims to explore the role of the lncRNA NEAT1/ mir-27b /Nrf2 signal axis in the development and treatment of ARDS/ALI in patients, as well as in LPS-induced ALI animal and cell models by using bioinformatics, molecular biology, histomorphology and clinical phenotype approaches, and to clarify the new mechanism in ARDS/ALI development and to provide new therapeutic targets.

DETAILED DESCRIPTION:
Collect blood and BALF from 400 ARDS patients at different time (at check-in, 24, 48 and 72 h after check-in the hospital) and 25 gender and age matching healthy controls. Use RT-PCR to detect the expression of lncRNA NEAT1、miR-27b and Nrf2 in blood and BALF of ARDS patients and health controls. The expressions of inflammatory and oxidative stress associated factors (NLRP3、NF-κB-P65、 p-P65、IκB、p-IκB、HO-1、NQO1、caspase-1、IL-1β、IL-6、IL-18、TNF-α) will be detected by western blot、ELISA and RT-PCR. Moreover, flow cytometry will be adopted to measure the numbers and kinds of cells in BALF. Then, analyze the differences of the expressions of lncRNA NEAT1、miR-27b and Nrf2 in the groups. To explore the correlation of expressions of lncRNA NEAT1、miR-27b and Nrf2 with inflammation and oxidative stress in the groups. Finally, to declare the relative of lncRNA NEAT1、miR-27b and Nrf2 with the time of mechanical ventilation, severity and mortality in 28 days of ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

We included patients with acute respiratory distress according to 2012 ARDS Berlin new definition (Acute Respiratory Distress Syndrome: The Berlin Definition. JAMA, 2012, 307(23):2526).

* Acute or progressive dyspnea within 1 week with identify cause;
* Chest radiograph/chest CT showed double lung infiltration, which could not be fully explained by pleural effusion, atelectasis, or nodules;
* Respiratory failure cannot be fully explained by heart failure and fluid overload;
* Hypoxemia, partial pressure of oxygen in arterial blood (PaO2)/oxygen fraction in air (FIO2) <150 mm Hg under PEEP ≥5 cm H2O, (mild ARDS: 200mmHg<PaO2/FiO2≤300mmHg, moderate ARDS: 100mmHg<PaO2/FiO2≤200mmHg, severe ARDS: PaO2/FiO2≤100mmHg);
* 18~70 years old;
* Agree to participate in the trial, and sign the informed consent.

Exclusion Criteria:

* Age less than 18 years old;
* Time of hospital stay <24 h;
* Pregnancy;
* Using V-V ECOM;
* Cardiac index <1.5L·ml.min-1.m-2;
* Pulmonary resection;
* Pulmonary embolism ;
* Refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We included ARDS patients from RICU、EICU、SICU、CCU in Beijing Anzhen hospital between 2020 and 2022
Sampling Method: Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The expression of lncRNA NEAT1 in blood and BALF in all groups | up to 24 day
  Use RT-PCR to measure the expression of lncRNA NEAT1 in blood and BALF in all groups
The expression of miR-27b in blood and BALF in all groups | up to 3 day
  Use RT-PCR to measure the expression of miR-27b in blood and BALF in all groups
The expression of Nrf2 in blood and BALF in all groups | up to 3 day
  Use RT-PCR and Wsetern blot to measure the expression of Nrf2 in blood and BALF in all groups
The expression of inflammatory factors(IL-1β、IL-6、IL-18、TNF-α) in blood and BALF in all groups | up to 3 day
  Use RT-PCR and ELISA to measure the expression of inflammatory factors(IL-1β、IL-6、IL-18、TNF-α) in blood and BALF in all groups
The expression of oxidative stress associated factors in blood and BALF in all groups | up to 3 day
  Use Western blot to measure the expression of oxidative stress associated factors(NLRP3、NF-κB-P65、 p-P65、IκB、p-IκB、HO-1、NQO1、caspase-1) in blood and BALF in all groups
The numbers and kinds of inflammatory cells in BALF and blood in all groups | up to 3 day
  Use flow cytometry to detect the number of inflammatory cells in BALF and blood in all groups
The kinds of inflammatory cells in BALF and blood in all groups | up to 3 day
  Use flow cytometry to detect the kinds of inflammatory cells(neutrophile、macrophage、 lymphocyte) in BALF and blood in all groups
The time of mechanical ventilation of patients in ARDS groups | up to28 day
  Record the time of mechanical ventilation of patients in ARDS groups
The severity of ARDS patients in ARDS groups | up to 28 day
  Record the severity(PaO2/FiO2、OI、S/F、OSI) of ARDS patients in ARDS groups
the mortality in 28 days of ARDS patients | up to 28 day
  Record the mortality in 28 days of ARDS patients

SECONDARY OUTCOMES:
The differences and correlation of the expressions of lncRNA NEAT1、miR-27b and Nrf2 in the groups | up to 28 day
  Analyse the differences of the expressions of lncRNA NEAT1、miR-27b and Nrf2 in the groups, and to explore the relations between the three(lncRNA NEAT1、miR-27b and Nrf2) in different groups.
The correlation of expressions of lncRNA NEAT1、miR-27b and Nrf2 with inflammation and oxidative stress in the groups. | up to 28 day
  To explore the correlation of expressions of lncRNA NEAT1、miR-27b and Nrf2 with inflammation and oxidative stress in the groups.
The relative of lncRNA NEAT1、miR-27b and Nrf2 with the time of mechanical ventilation, severity and mortality in 28 days of ARDS patients | up to 28 day
  To declare the relative of lncRNA NEAT1、miR-27b and Nrf2 with the time of mechanical ventilation, severity and mortality in 28 days of ARDS patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Respiratory and Critical Care Medicine, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart, Lung and Blood Vessel Diseases, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Fan E, Brodie D, Slutsky AS. Acute Respiratory Distress Syndrome: Advances in Diagnosis and Treatment. JAMA. 2018 Feb 20;319(7):698-710. doi: 10.1001/jama.2017.21907. PMID 29466596
- [Background] Lu MC, Ji JA, Jiang ZY, You QD. The Keap1-Nrf2-ARE Pathway As a Potential Preventive and Therapeutic Target: An Update. Med Res Rev. 2016 Sep;36(5):924-63. doi: 10.1002/med.21396. Epub 2016 May 18. PMID 27192495
- [Background] Wei J, Chen G, Shi X, Zhou H, Liu M, Chen Y, Feng D, Zhang P, Wu L, Lv X. Nrf2 activation protects against intratracheal LPS induced mouse/murine acute respiratory distress syndrome by regulating macrophage polarization. Biochem Biophys Res Commun. 2018 Jun 7;500(3):790-796. doi: 10.1016/j.bbrc.2018.04.161. Epub 2018 Apr 25. PMID 29684352
- [Background] Liu Q, Lv H, Wen Z, Ci X, Peng L. Isoliquiritigenin Activates Nuclear Factor Erythroid-2 Related Factor 2 to Suppress the NOD-Like Receptor Protein 3 Inflammasome and Inhibits the NF-kappaB Pathway in Macrophages and in Acute Lung Injury. Front Immunol. 2017 Nov 9;8:1518. doi: 10.3389/fimmu.2017.01518. eCollection 2017. PMID 29163554
- [Background] Liu Y, Song M, Zhu G, Xi X, Li K, Wu C, Huang L. Corynoline attenuates LPS-induced acute lung injury in mice by activating Nrf2. Int Immunopharmacol. 2017 Jul;48:96-101. doi: 10.1016/j.intimp.2017.04.029. Epub 2017 May 6. PMID 28486213
- [Background] Rajasekaran S, Pattarayan D, Rajaguru P, Sudhakar Gandhi PS, Thimmulappa RK. MicroRNA Regulation of Acute Lung Injury and Acute Respiratory Distress Syndrome. J Cell Physiol. 2016 Oct;231(10):2097-106. doi: 10.1002/jcp.25316. Epub 2016 Feb 4. PMID 26790856
- [Background] Wu CT, Huang Y, Pei ZY, Xi X, Zhu GF. MicroRNA-326 aggravates acute lung injury in septic shock by mediating the NF-kappaB signaling pathway. Int J Biochem Cell Biol. 2018 Aug;101:1-11. doi: 10.1016/j.biocel.2018.04.019. Epub 2018 May 1. PMID 29727715 (Retraction: PMID 33516658 Int J Biochem Cell Biol. 2021 Mar;132:105922)
- [Background] Ling Y, Li ZZ, Zhang JF, Zheng XW, Lei ZQ, Chen RY, Feng JH. RETRACTED: MicroRNA-494 inhibition alleviates acute lung injury through Nrf2 signaling pathway via NQO1 in sepsis-associated acute respiratory distress syndrome. Life Sci. 2018 Oct 1;210:1-8. doi: 10.1016/j.lfs.2018.08.037. Epub 2018 Aug 17. PMID 30121199
- [Background] Ding L, Ni J, Yang F, Huang L, Deng H, Wu Y, Ding X, Tang J. Promising therapeutic role of miR-27b in tumor. Tumour Biol. 2017 Mar;39(3):1010428317691657. doi: 10.1177/1010428317691657. PMID 28351320
- [Background] Zhou R, Gong AY, Eischeid AN, Chen XM. miR-27b targets KSRP to coordinate TLR4-mediated epithelial defense against Cryptosporidium parvum infection. PLoS Pathog. 2012;8(5):e1002702. doi: 10.1371/journal.ppat.1002702. Epub 2012 May 17. PMID 22615562
- [Background] Signorelli SS, Volsi GL, Pitruzzella A, Fiore V, Mangiafico M, Vanella L, Parenti R, Rizzo M, Volti GL. Circulating miR-130a, miR-27b, and miR-210 in Patients With Peripheral Artery Disease and Their Potential Relationship With Oxidative Stress. Angiology. 2016 Nov;67(10):945-950. doi: 10.1177/0003319716638242. Epub 2016 Jul 11. PMID 26980776
- [Background] Li T, Cao H, Zhuang J, Wan J, Guan M, Yu B, Li X, Zhang W. Identification of miR-130a, miR-27b and miR-210 as serum biomarkers for atherosclerosis obliterans. Clin Chim Acta. 2011 Jan 14;412(1-2):66-70. doi: 10.1016/j.cca.2010.09.029. Epub 2010 Sep 29. PMID 20888330
- [Background] Huang Y, Huang L, Zhu G, Pei Z, Zhang W. Downregulated microRNA-27b attenuates lipopolysaccharide-induced acute lung injury via activation of NF-E2-related factor 2 and inhibition of nuclear factor kappaB signaling pathway. J Cell Physiol. 2019 May;234(5):6023-6032. doi: 10.1002/jcp.27187. Epub 2018 Dec 24. PMID 30584668
- [Background] Song YX, Sun JX, Zhao JH, Yang YC, Shi JX, Wu ZH, Chen XW, Gao P, Miao ZF, Wang ZN. Non-coding RNAs participate in the regulatory network of CLDN4 via ceRNA mediated miRNA evasion. Nat Commun. 2017 Aug 18;8(1):289. doi: 10.1038/s41467-017-00304-1. PMID 28819095
- [Background] Yan B, Yao J, Liu JY, Li XM, Wang XQ, Li YJ, Tao ZF, Song YC, Chen Q, Jiang Q. lncRNA-MIAT regulates microvascular dysfunction by functioning as a competing endogenous RNA. Circ Res. 2015 Mar 27;116(7):1143-56. doi: 10.1161/CIRCRESAHA.116.305510. Epub 2015 Jan 13. PMID 25587098
- [Background] Wang Y, Xu Z, Jiang J, Xu C, Kang J, Xiao L, Wu M, Xiong J, Guo X, Liu H. Endogenous miRNA sponge lincRNA-RoR regulates Oct4, Nanog, and Sox2 in human embryonic stem cell self-renewal. Dev Cell. 2013 Apr 15;25(1):69-80. doi: 10.1016/j.devcel.2013.03.002. Epub 2013 Mar 28. PMID 23541921
- [Background] Xiong DD, Li ZY, Liang L, He RQ, Ma FC, Luo DZ, Hu XH, Chen G. The LncRNA NEAT1 Accelerates Lung Adenocarcinoma Deterioration and Binds to Mir-193a-3p as a Competitive Endogenous RNA. Cell Physiol Biochem. 2018;48(3):905-918. doi: 10.1159/000491958. Epub 2018 Jul 23. PMID 30036873
- [Background] Wang L, Xia JW, Ke ZP, Zhang BH. Blockade of NEAT1 represses inflammation response and lipid uptake via modulating miR-342-3p in human macrophages THP-1 cells. J Cell Physiol. 2019 Apr;234(4):5319-5326. doi: 10.1002/jcp.27340. Epub 2018 Sep 27. PMID 30259979